CLINICAL TRIAL: NCT05201781
Title: Long-term Follow-up Study for Participants Previously Treated With Ciltacabtagene Autoleucel
Brief Title: A Long-term Study for Participants Previously Treated With Ciltacabtagene Autoleucel
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR109123; 68284528MMY4002 (Other: Janssen Research & Development, LLC); 2020-005521-84 (EudraCT Number); 2023-505530-10-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05346835 (Available)
Record Dates: First submitted 2022-01-10; First posted 2022-01-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cilta-cel (Experimental): Participants who had previously received treatment with cilta-cel in a Company-sponsored clinical study (example, NCT04923893, NCT03758417, NCT04181827, NCT05347485, NCT04133636, and NCT03548207) in the global development program will be enrolled into this study once the individual's participation in the particular interventional study has ended or a study has been terminated. Participants will not receive any treatment in this study and will be followed-up at least once per year on delayed adverse events for up to 15 years after receiving the last dose of cilta-cel.
  Interventions: Drug: Cilta-cel

INTERVENTIONS:
Drug: Cilta-cel — Participants who had received cilta-cel in previous studies will be followed up in this study. No additional study treatment will be administered to participants in this study.
  Other Names: JNJ-68284528; LCAR-B38M CAR-T cells

SUMMARY:
The purpose of this study is to collect long-term follow-up data on delayed adverse events after administration of ciltacabtagene autoleucel (cilta-cel), and to characterize and understand the long-term safety profile of cilta-cel.

DETAILED DESCRIPTION:
Cilta-cel (JNJ-68284528/LCAR-B38M chimeric antigen receptor T-cells [CAR-T]) is an autologous CAR-T therapy that targets B-cell maturation antigen (BCMA), a molecule expressed on the surface of mature B lymphocytes and malignant plasma cells. There will be no treatment administered during the study and the data obtained from this study will help to assess whether there will be long-term cilta-cel-related toxicities. The study will consist of 2 phases: within the first 5 years after receiving the last dose of cilta-cel and Year 6 to 15 years after last dose of cilta-cel. Safety evaluations will include a review of adverse events, laboratory test results, and physical examination findings (including neurological examination). The duration of the study is up to 15 years after last dose of cilta-cel and participants will be followed at least once per year.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have received at least one dose of cilta-cel in a Company-sponsored clinical study
* Participants who have provided informed consent for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2037-07-29 (Estimated); Study Completion 2037-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with New Malignancies and Recurrence of Pre-existing Malignancy | Up to 15 years
  Number of participants with new malignancies and recurrence of pre-existing malignancy will be reported.
Number of Participants with New Incidence or Exacerbation of a Pre-existing Neurologic Disorder | Up to 15 years
  Number of participants with new incidence or exacerbation of a pre-existing neurologic disorder will be reported.
Number of Participants with New Incidence or Exacerbation of a Pre-existing Rheumatologic or Other Autoimmune Disorder | Up to 15 years
  Number of participants with new incidence or exacerbation of a pre-existing rheumatologic or other autoimmune disorder will be reported.
Number of Participants with New Incidence of Grade Greater than or Equal to (>=) 3 Hematologic Disorder Including Hypogammaglobulinemia | From year 1 up to year 5
  Number of participants with new incidence of Grade >=3 hematologic disorder including hypogammaglobulinemia will be reported.
Number of Participants with Serious Hematologic Disorder, including Hypogammaglobulinemia | From year 6 up to year 15
  Number of participants with serious hematologic disorder, including hypogammaglobulinemia will be reported. Serious hematologic disorder, includes hypogammaglobulinemia (all grades, regardless of causality).
Number of Participants with New Incidence of Grade >= 3 Infection | From year 1 up to year 5
  Number of participants with new incidence of Grade >=3 infection will be reported.
Number of Participants with Serious Infection | From year 6 up to year 15
  Number of participants with serious infection will be reported. Serious infection includes all grades, regardless of causality.
Number of Participants with Serious Adverse Events (SAEs) | From year 1 up to year 5
  A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Number of Participants with Related Serious Adverse Events Assessed by the Investigator | From year 6 up to year 15
  Number of participants with related serious adverse events assessed by the investigator will be reported. A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.

SECONDARY OUTCOMES:
Number of Participants with Measurable Replication Competent Lentivirus (RCL) in Peripheral Blood | Up to 15 years
  Number of participants with measurable RCL in peripheral blood will be reported.
Number of Participants with Chimeric Antigen Receptor (CAR) Transgene Level Greater Than (>) Lower Limit of Quantitation (LLOQ) in Peripheral Blood Cells | Up to 15 years
  Number of participants with CAR transgene level >LLOQ in peripheral blood cells will be reported.
Pattern of Lentiviral Vector Integration Sites | Up to 15 years
  Pattern of lentiviral vector integration sites if at least 1 percent (%) of cells in the blood sample or new malignancy are positive for vector sequences will be reported.
Investigator's Response Assessment of Long Term Follow-up on Chimeric Antigen Receptor T-cell (CAR-T) Therapy Based on Local Lab Assessments | Up to 15 years
  Investigator's response assessment of long term follow-up on CAR-T therapy based on local lab assessments if the participant does not have confirmed disease progression or does not initiate subsequent anti-myeloma therapy at the entry of the study and at any time of during the study will be reported.
Overall Survival (OS) | Up to 15 years
  OS is measured from the date of randomization to the date of the participant's death.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (50):
- United States (28):
  - Mayo Clinic Cancer Center-Scottsdale, Phoenix, Arizona
  - City of Hope, Duarte, California
  - University of California San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Kansas University Medical Center, Westwood, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School Of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Froedtert Memorial, Milwaukee, Wisconsin
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- China (11):
  - Peking University Third Hospital, Beijing
  - West China Hospital Si Chuan University, Chengdu
  - Fujian Medical University Union Hospital, Fuzhou
  - Sun Yat-sen University Cancer Hospital, Guangzhou
  - First Hospital, Zhejiang University Medical College, Hangzhou
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - Shanghai Changzheng Hospital, Shanghai
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
  - Shanghai Fourth People s Hospital, Shanghai
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
- France (2):
  - CHRU de Lille Hopital Claude Huriez, Nord
  - Hopital Saint Louis, Paris
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Japan (2):
  - Nagoya City University Hospital, Nagoya
  - Japanese Red Cross Medical Center, Shibuya City
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam
  - University Medical Center Groningen, Groningen
- Spain (2):
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency